CLINICAL TRIAL: NCT04208295
Title: 24-hour Blood Pressure Dynamics and Autonomic Adrenergic Regulation in Type 2 Diabetics
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Other Study IDs: IDNC_Adrenergic_BP_Testing
Record Dates: First submitted 2019-12-19; First posted 2019-12-23 (Actual); Last update posted 2019-12-23 (Actual); Status verified 2019-05

CONDITIONS: Diabetes Mellitus, Type 2; Polyneuropathy Diabetes; Autonomic Neuropathy; Diabetic Neuropathies; Diabetic Complications Neurological
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetic Neuropathies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients: Type 2 diabetics
- Healthy controls: Matched healthy controls

SUMMARY:
Autonomic neuropathy is a common complication of type 2 diabetes mellitus. Symptoms from cardiovascular autonomic neuropathy include, dizziness, orthostatic hypotension and insufficient heart rate and blood pressure (BP) regulation during physical exertion. The degree of cardiovascular autonomic neuropathy is most commonly measured as cardiac autonomic neuropathy based on at least two abnormal cardiac reflex tests, which primarily measures parasympathetic indices of the autonomic nervous system (ANS).

Few measures are available for quantifying the sympathetic/adrenergic branch of the ANS.

Circadian changes in BP is a documented measure of BP variability, regulated centrally by a multitude of centers. A growing number of studies indicate that a diminished BP variability is associated with increased cardiovascular risk and injury. The ANS plays a pivotal role in the execution of these circadian BP changes, mainly through sympathetic adrenergic nerve fibers

Few studies have investigated the applicability of 24-hour indices as predictor for autonomic adrenergic dysfunction. No previous studies have investigated the association between clinical markers of adrenergic function, and 24-hour blood pressure indices in type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes
* Normal 12-lead ECG

Exclusion Criteria:

* Significant cardiovascular, muscular, lung, kidney or psychiatric disease
* Pregnancy
* Malignant disease, HIV, alcoholism or drug abuse
* Parkinson disease
* Ischemic heart disease
* Vital medicine that can affect the autonomic nervous system

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Type 2 diabetics previously screened for diabetic polyneuropathy will be invited
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2019-05-01 (Actual); Primary Completion 2020-06 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
24 hour Blood Pressure | 0
  Day/night blood pressure ratio. Day time standard deviation and average real time variation
Autonomic adrenergic measure | 0
  Valsalva maneuver - Phase 2Late, Pressure recovery time, Baroreceptor sensitivity, Phase 4 rise. Head up tilt test - Blood pressure dip ratio

CONTACTS AND LOCATIONS:
Locations (1):
- Danish Pain Research Center, Aarhus University Hospital, Aarhus, Skejby, Denmark